CLINICAL TRIAL: NCT04312516
Title: Addenbrooke's Cognitive Examination III Scale as a Screening Tool for Cognitive Impairment in Surgical Population: Validity and Reliability of the Culturally Adapted Greek Version
Brief Title: Greek Validation of ACE III Test in Perioperative Patients
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Maria Zouka, Consultant - Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: ACEIIIPREOP
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: ACE III; MoCA; Neurocognitive dysfunction; Perioperative
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Participants scheduled for surgery with MoCA score ≥ 26 preoperatively
- Patients: Participants scheduled for surgery with MoCA score < 26 preoperatively

SUMMARY:
Postoperative neurocognitive disorders, including postoperative delirium (POD) and postoperaive cognitive dysfunction (POCD), are common complications of perioperative neurocognition in elderly patients undergoing surgery. POD and POCD have short- and long-term consequences, such as increased hospital stays and costs, augmented morbidity and mortality, as well as higher risk for cognitive decline later in life. Therefore, early prevention and diagnosis of these conditions is of great importance.

A number of psychometric tests have been proposed as cognitive screening tools. Given the fact that many of them show weaknesses and difficulties in performance, scientists have sought for more useful alternatives. Montreal Cognitive Assessment (MoCA) is considered to be a good choice, as it has been successfully applied in the perioperative setting. What's more, it has been translated and validated for a Greek population with neurological disorders. Addenbrooke's Congnitive Examination III (ACE III) has been introduced recently into clinical practice. It is an easy to perform and detailed test that covers several neurocognitive domains and has shown high sensitivity and specificity in clinical conditions, including dementia and Alzheimer's disease. Although current literature lacks data concerning its perioperative use, ACE III could prove useful for screening patients undergoing surgery and anesthesia on the basis of its favorable characteristics as mentioned above.

The aim of this study is to translate the ACE III (English version 2012) into Greek and assess its validity in perioperative patients aged >55 years.

DETAILED DESCRIPTION:
In this prospective cohort study, the ACE III will be translated and adapted into the Greek language by the researchers according to the relative guidelines for cultural adaptation. Backward translation will be performed by a fluent bilingual specialist to ensure the optimum reliability of the questionnaire.

A total of 128 surgical patients are planned to be enrolled in the study protocol after informed consent. Primary screening of the whole population will be conducted at the pre-admission clinic using the MoCA test by two examiners in order to determine their cognitive status. Simultaneously, the ACE III will be applied to set the baseline measurements for each participant. Subjects with MoCA score <26 will form the patients' group while those with MoCA scores at least 26 will form the control group.

Screening with both MoCA and ACE-III tests will be repeated the day before surgery with at least a 7-day gap between the two assessments.

Total scores and subscores at both time-points will be calculated and comparative performance of all participants will be assessed after statistical analysis of collected data.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgical intervention
* At least of primary level of education

Exclusion Criteria:

* Neurodegenerative disease
* Cerebrovascular disease
* Psychiatric disorders
* History of head injury
* Use of medication affecting the CNS

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 128 surgical patients (cognitively and non-cognitively impaired)
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Cultural adaption | 2 months
  Cultural adaption of ACE III (English version 2012) into the Greek language
Validation | 2 months
  Construct and convergent validity of the translated version of ACE III into the Greek language

CONTACTS AND LOCATIONS:
Overall Officials: Maria Zouka, MD, Principal Investigator — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No